CLINICAL TRIAL: NCT05223322
Title: DECODE Heartland: Understanding and Addressing Disparities in Cancer Therapy Induced Inflammation and Associated Endothelial Dysfunction
Brief Title: Understanding and Addressing Disparities in Cancer Therapy Induced Inflammation and Associated Endothelial Dysfunction
Acronym: DECODE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Melinda Stolley, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00041443
Record Dates: First submitted 2021-11-16; First posted 2022-02-03 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Thrombin Time; Methods

STUDY DESIGN:
Masking Description: Following baseline data collection, participants will be randomized into one of two study arms: intervention (exercise) and control (usual care). The investigators have three strata in this study: 1) race/ethnicity (NHW or Bl/AA), 2) anti-cancer therapy (ANTs, anti-Her2 treatments, or both), and 3) comorbidity profile (low vs. high). (High comorbidity level is defined as >3 comorbidities that include hypertension, diabetes, hyperlipidemia, BMI 50+, renal failure, liver failure. It is possible there may be other comorbidities that may be identified based on physician feedback and patient approval). The investigators will employ blocked randomization within each site (MCW and UIC) that have their own stratified randomization sequence. Each patient will be randomized to a treatment arm (usual care or exercise) via MCW's OnCore Clinical Trials Management System at the MCW Clinical Trials Office.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Taking Charge during Treatment (TCT) Intervention (Active Comparator): Taking Charge during Treatment (TCT) Intervention. TCT is a 16-20week intervention that promotes adoption of the ACSM exercise guidelines for cancer survivors during treatment, including regular moderate to vigorous physical activity (150 minutes per week of moderate activity or 75 minutes per week of vigorous activity) and a minimum of twice weekly resistance training (RT) minutes during CTx and after. Participants will receive "Take Charge" program binder, 2-4 x weekly text messaging, activity tracker and resistance bands.
  Interventions: Behavioral: Taking Charge during Treatment (TCT) Intervention
- Control Group (No Intervention): To ensure scientific rigor allowing us to test causal pathways associated with exercise, women will be randomized to the TCT intervention or control group arm. The control group will not receive the TCT intervention The investigators experience teaches us that to increase the likelihood of retaining control group participants, the investigators must offer some resources. Thus, the investigators will provide the control group with a one-page summary of the American College of Sports Medicine exercise recommendations, and the "Take Charge" program binder at the completion of the study. Participants will also receive resistance bands and activity tracker at the end of the study. 95 The investigators will also send weekly text messages with supportive content not related to exercise or lifestyle (i.e., a riddle, "take a moment to smile today," a picture of a baby animal).

INTERVENTIONS:
Behavioral: Taking Charge during Treatment (TCT) Intervention — CT is a 16-20week intervention that promotes adoption of the ACSM exercise guidelines for cancer survivors during treatment, including regular moderate to vigorous physical activity (150 minutes per week of moderate activity or 75 minutes per week of vigorous activity) and a minimum of twice weekly resistance training (RT) minutes during CTx and after. Program components include (1) a binder of information, (2) weekly coaching, (3) 2-4x weekly text messaging and (4) exercise supplies. The TCT program is grounded in Social Cognitive Theory.
  Arms: Taking Charge during Treatment (TCT) Intervention

SUMMARY:
Very little is understood about the off-target vascular mechanisms of anti-cancer drug toxicity and the impact of exercise on these changes. Much of what has been learned about molecular pathways regulating vascular endothelial function has been established by logical expansion of knowledge obtained through experimental studies (e.g., discovery of endothelium-derived relaxing factor/nitric oxide). Within the last 10 years technological advancements of -omics approaches, such as RNA-sequencing and shotgun proteomics, have dramatically reduced the cost and technical challenge of accessing these tools for discovery-based research. Investigators are now able to obtain unbiased datasets showing changes in transcript or protein expression within complex samples. With cost and accessibility of sequencing is no longer being substantial bottleneck, one of major challenges researchers now face is determining how to meaningfully interpret profiles from large datasets. The extensive characterization of molecular pathways impacting inflammatory responses, endothelial function and angiogenesis, the pathway and network analysis tools will be an asset for identification molecular pathways relevant to alterations in microvascular endothelial function. The investigators preliminary studies on only a small number of samples highlights this potential of the proposed approach to lead to identify personalized medicine-based profiles that will predict patients are likely to develop microvascular endothelial dysfunction from CTx.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) assigned female sex at birth
* Diagnosed with invasive non-metastatic breast cancer
* Receiving neo-adjuvant CTx (or adjuvant CTx and undergoing breast conserving surgery) that includes anthracyclines (such as DOX) and/or targeted anti-Her2 therapy
* Able to safely participate in moderate exercise and strength training based on MD approval
* Willing to complete all study activities
* Self-identifies as Black/African American or non-Hispanic White

Exclusion Criteria:

* Unintentional weight loss > 10% in the past 6 months
* Current pregnant and lactating patients. Must have completed lactation prior to study start
* Metastatic disease
* Diagnosed cardiovascular disease as evidenced by cardiomyopathy (reduced regional or global LV contractility), diastolic dysfunction grade 2 or above, symptomatic coronary - artery disease, ejection fraction below 50%
* History of prior chemotherapy or targeted H2N Treatment received less than 3 years ago
* Non-English speaking

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females currently diagnosed with Breast Cancer
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximal Exercise: Maximal oxygen consumption will be evaluated using cycle ergometry or treadmill to exhaustion as described in the Integrative Physiology Laboratory at each testing visit. | T1 (baseline), T2 (18-24 weeks), and T3 (12 months)
  Investigators will use a graded protocol, starting at 50 watts followed by 30 watt increments every 2 minutes. Subjects will be connected to a breath-by-breath metabolic system (Cosmed, Italy) for measurement of VO2peak. A maximal effort will be defined as fulfillment of three of the following criteria: 1) A plateau in VO2 with an increase in work rate defined as an increase in VO2 of less than 50 ml/min; 2) A maximal HR within 10 beats of predicted maximal heart rate; 3) A respiratory exchange ratio of greater than 1.15; 4) No increase in heart rate with an increase in work rate (less than 3 beats); or 5) A rating of perceived exertion of 18 or greater on the Borg scale. These criteria are according to and consistent with the AHA exercise testing guidelines and performed regularly in Dr. Phillips' and Dr. Durand's laboratory groups59, 62-66.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - General (FACT-B) | T1 (baseline), T2 (18-24 weeks), and T3 (12 months)
  This survey measures physical, social, emotional, and functional wellbeing and wellness and symptoms associated with breast cancer and its treatments.
The Distress Thermometer | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  This is a simple tool to effectively screen for symptoms of distress.
Perceived Stress Scale | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  This survey is a class stress assessment to help understand how different situations affect feelings and perceived stress, asking about thoughts and feelings.
Hospital Anxiety and Depression Scale | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  This will measure anxiety and depression in a general medical population of patients.
The Functional Assessment of Chronic Illness Therapy - Fatigue | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  Participants will self-report fatigue and its impact upon daily activities and function.
PROMIS - Social Support | T1 (baseline), T2 (18-40 weeks), and T3 (12 months)
  This survey will assess how much social support each individual has in their personal network.
PROMIS - Pain Interference | T1 (baseline), T2 (18-24 weeks), and T3 (12-15 months)
  This instrument will measure the self-reported consequences of pain on relevant aspects of a person's life.
Assess mitochondrial DNA damage | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  Mitochondrial DNA damage will be assessed in isolated vessels from biopsies and total peripheral blood mononuclear blood cells (PBMCs) via a well-established PCR protocol. Similarly, a PCR based method is used to quantify levels of cell free mtDNA in plasma samples from study participants.
Cytokine analysis | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  Investigators will utilize Isoplex platform via CodePlex Human Cytokine Storm Panel-8 to quantify a large array of inflammatory cytokines using minimal amounts (<30 ul) of plasma sample.
Gene Express Profiling | T1 (baseline), T2 (18-40 weeks), and T3 (115 months)
  Transcriptomic expression profiling of PBMC and endothelial cells will be performed utilizing existing infrastructure (Genomic Sciences and Precision Medicine Center at MCW). RNA sequencing will be performed Illumina on NovaSeq sequencer.
Endothelial function | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  Microvascular function from gluteal and surgical fat biopsies will be used to test the direct effect of clinically used chemotherapy on peripheral microvascular function (as surrogate for coronary microvessels). Investigators propose to perform studies before, after the chemotherapy regimen, and at 12 months follow up. Study team evaluate microvascular dilator capacity, both endothelial and smooth muscle mediated, and quantify levels of vasodilators (NO and H2O2) via fluorescent probes.
Flow Mediated Dilation | T1 (baseline), T2 (18-40 weeks), and T3 (12 months)
  Flow mediated dilation of the brachial artery (large conduit vessels) will be assessed using ultrasound in a noninvasive manner.
Cardiac function - Echocardiagram | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  Echocardiograms: Aortic diameter, cardiac output, stroke volume, heart rate, end diastolic, and end systolic volume will be assessed at rest using two-dimensional echocardiography. With subjects in the left lateral position, measurements will be obtained using the two (Parasternal and Short Axis) and four-chamber view.
Cardiac function - Pulse Wave Velocity | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  Pulse Wave Velocity: A non-invasive technique will be used to measure arterial stiffness (pulse wave velocity and central pressures). Briefly, investigators will record waveforms at the carotid and femoral arteries using tonometry and a partially inflated pressure cuff placed over the upper arm and thigh. The distance between sites will be determined using a tape measure.
Cognitive Function | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  PROMIS - Cognitive Function Short Form: This is a short six-item sub-set scale of the full PROMIS Cognitive Function item bank that assesses patient-perceived cognitive deficits

OTHER OUTCOMES:
DEXA Scan | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  Body composition: DXA imaging is a 10 minute, noninvasive, technique that provides precise whole-body measurements of fat (total and visceral) and lean mass. Certified DXA technologists will perform and analyze whole body measures using the same machine for each participant at each time point. To ensure reliability and precision, machines are calibrated daily.
Height and Weight | T1 (baseline), T2 (18-24 weeks), and T3 (12-15 months)
  Height and Weight: To calculate BMI, investigators will will assess height (baseline only) using a portable stadiometer and weight using a digital scale with participants wearing light clothes and no shoes. A 0.2 kg discrepancy in weight or a 0.5 cm discrepancy in height in the first two measurements, will result in a third measurement.
Accelerometry | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  Accelerometry. Summary measures of PA levels will be derived from 7-day accelerometer wear data (% time sedentary, % time moderate to vigorous PA, counts per minute). Study team will adopt the common guideline of 10 hours or more of wear time necessary to define a valid day. Investigators will use the Troiano cut points (sedentary, light, moderate, vigorous).
Physical Activity self report | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  Godin Leisure Activity Index collects data on mild, moderate, and vigorous activity.
Pittsburgh Sleep Quality Index | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  This is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas.
Sitting Time Questionnaire | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  The STQ is a 5-question self-report survey asking about amount of time spent sedentary.
Handgrip strength | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  Measured with a Takei handgrip dynamometer. This test of LM function correlates with total body muscle strength73 and mortality74.
Sit to Stand | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  Number of completed Sit to Stand repetitions performed in 30 secs using a chair with no arms with a height of approximately 43 cm75.
6 Minute Walk Test | T1 (baseline), T2 (18-40 weeks), and T3 (12-15 months)
  Total distance traveled in 6 mins is recorded and used to determine endurance.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Illinois Chicago, Chicago, Illinois
  - Medical College of Wisconsin, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided